CLINICAL TRIAL: NCT07384650
Title: Post-discharge Nurse-led Rehabilitation to Improve Functional Activity and Community Participation Among Stroke-Patients in Bangladesh: A Randomized Controlled Trial
Brief Title: Post-stroke Nurse-led Rehabilitation to Improve Functional Activity and Community Participation in Bangladesh
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hiroshima University (Other)
Responsible Party: Principal Investigator, Salma Akhter, Principal Investigator, Hiroshima University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRB/NINS/2025/535
Record Dates: First submitted 2026-01-25; First posted 2026-02-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Stroke
Keywords: Stroke; rehabilitation; functional activity; participation
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Participants will be trained in self-care with stroke disabilities (e.g. eating, grooming, bathing, dressing, toileting), physical exercise, lifestyle modification, prevention of complications after stroke through researcher developed "Health booklet". Based on their disabilities, some assistive and exercise devices will be provided to them for improving functional independence.
  After discharge they will be educated and followed by RA nurses through tele services for 6 months. The nurses will contact the participants periodically over the telephone, and follow up on their regular self-care activities, adjustment to devices, exercise and participatory behavior.
  Interventions: Device: in daily everyday routine practice
- Control Group (No Intervention): The participants in CG will not receive "Education booklet" or assistive device . They will receive the usual rehabilitation education from the hospital.

INTERVENTIONS:
Device: in daily everyday routine practice — Participants will be provided with education booklet and assistive devices for implement in their daily life to improve their functional activity.
  Other Names: Education Booklet
  Arms: Intervention Group

SUMMARY:
Stroke causes various levels of disability which decreases physical function for a prolonged period. The purpose of this study is to evaluate the effectiveness of a nurse-led rehabilitation program including a multidisciplinary team focused on improving the functional ability among post-stroke patients in Bangladesh. A prospective, open-label (1:1) randomized controlled trial (RCT) will be conducted at the National Institute of Neuroscience & Hospital (NINS&H) in Dhaka, Bangladesh from January 2026 to September 2026. Participants will be the post-stroke patients who got discharged from NINS&H within 2 weeks after the onset of stroke and the family caregivers of the patients and meet the inclusion criteria. The sample size will be calculated based on G-Power analysis with a medium effect size and will be 166. The intervention will be designed to provide the 6-months Nurse-led rehabilitation program including a multidisciplinary team regarding self-care and the use of assistive devices. Assessment for rehabilitation will be performed by the multidisciplinary team with research nurses (RA nurses), physiotherapists (PT) and occupational therapists (OT). The control group will receive the usual care. The primary outcome is improved activity and participation measured by the Functional Independence Measurement (FIM). The secondary outcomes are improved motor function, self-efficacy, emotional status and participation ability. The endpoints will be compared at baseline, 3rd and 6th months. We assume that patients receiving rehabilitation education and assistive device progress to achieve an optimal level of independence, with improved motor function, emotional status and participation ability to re-integrate into society.

DETAILED DESCRIPTION:
Stroke is a significant cause of adult death and disability globally, leading to clinical, social, and economic challenges for individuals, families, and healthcare systems. Over 12 million new strokes are reported each year, with about 50% of survivors facing long-term functional impairments that affect their ability to live independently [1]. Post-acute disability commonly comprises motor deficits, cognitive and perceptual dysfunction, communication disorders, and restrictions in activities of daily living (ADLs), greatly diminishing quality of life [2]. Consequently, rehabilitation is essential in stroke management to restore function, avert complications, and support community reintegration [3].

Growing evidence indicates that stroke rehabilitation is most effective with a multidisciplinary team (MDT) model, incorporating physiotherapists, occupational therapists, speech-language pathologists, rehabilitation physicians, psychologists, and nurses [4]. MDT-based rehabilitation facilitates coordinated goal setting, individualized therapy plans, and early identification of barriers to progress [5]. When compared to non-coordinated care, systematic studies and clinical guidelines consistently show that planned and interdisciplinary stroke care improves functional outcomes, lowers mortality, and increases the chance of returning home after stroke [6, 7].

Post-acute rehabilitation, following medical stabilization, is vital for enhancing neuroplasticity as targeted interventions during this phase can improve motor function, cognitive function, and functional independence [8]. Patients receiving intensive post-acute therapy exhibited significantly better gains in mobility, self-care, and participation outcomes over 12 weeks compared to lower-intensity groups [9]. Studies found that combining cognitive-motor therapy with traditional MDT practice improved executive function and ADL performance across a 6-week period. These findings underscore the value of holistic MDT programs in addressing the multidimensional impairments common in stroke survivors [10].

Adherence to rehabilitation is a behavior that indicates the patient's commitment to and willingness to engage in the planned therapy regimen and treatment to improve daily living activities, quality of life, and outcomes as well as prevent complications and recurrence of stroke [11, 12]. Treating chronic illnesses like stroke, adherence to long-term therapies, particularly rehabilitation, is a significant healthcare challenge [13]. Digital health approaches like tele-services with personalized advice, emotional support, and time influences for enhancing rehabilitation adherence in stroke patients as relevant quality feedback significantly improves adherence [14]. Medical experts emphasize that key determinants of adherence in out-of-hospital rehabilitation include access to tele-rehabilitation, tele-medical resources, and active participation from outpatient clinics highlighting the need for attention to both in- and out-of-hospital rehabilitation [15]. For effective rehabilitation, a reliable scale to measure patient adherence to the regimen is essential.

Nurse-led rehabilitation and care for stroke patients combined with a multidisciplinary team significantly improves motor recovery, functional independence (ADL), and quality of life and self-management when compared to standard care [16]. Acute care, rehabilitation, discharge, and community/home-based follow-up can all be bridged by nurse-led programs, which are typically feasible, effective, and acceptable [17].

In LMICs including Bangladesh, there is a lack of institutional acute, post-acute and long-term rehabilitation services available after receiving acute care management from the hospital [18]. Patients with disabilities who need rehabilitation suffer due to inadequate healthcare infrastructure and financial resources [19]. As there are insufficient post-stroke institutional services available in Bangladesh, home-based stroke rehabilitation could be an alternative way to play a vital role in ensuring continuity of care and supporting functional recovery within patients' home environments [20].

Therefore, this study will explore the effectiveness of a structured nurse-led multidisciplinary post-acute rehabilitation program. This study would provide more rigorous evidence on whether coordinated, team-based rehabilitative interventions significantly enhance functional independence compared to conventional rehabilitation approaches in Bangladesh. The findings could guide clinical practice standards, support the development of optimized rehabilitation pathways for stroke survivors and reform health-care policy for the disabled.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years old and above, both males & females,
2. Irrespective of the type of stroke and time of stroke,
3. mRS 2-4 with disability on upper and/or lower limb(s)
4. Physician advice on rehabilitation, and who needs assistive devices for ADL,
5. Having a phone, and
6. Willing to provide consent & participate in the study.

Exclusion Criteria:

1. Participation in other clinical trials,
2. Planning to receive institutional rehabilitation services, and
3. Cannot communicate (having speech difficulties).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Estimated)
Dates: Start 2026-01-30 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Improved Functional Activity | 6 months
  It will be measured by Functional Independence Measurement (FIM). The FIM was developed in 1983 by a task force from the American Congress of Rehabilitation Medicine (ACRM) and the American Academy of Physical Medicine and Rehabilitation (AAPM&R) [23]. The Bengali version of the scale was implemented among the functionally disabled patients in Bangladesh and found to be valid and reliable (α = 0.97) [24]. This scale has 18 items from level 1-total assistance to level 7-complete independence. This scale consists of 2 sub-scales including physical (13 items) and cognitive (5 items) domains. The physical domain score ranges from 13-91 and the cognitive domain score ranges from 5-35. The total score range is from 18-126. The higher the score, the better the level of independence.

SECONDARY OUTCOMES:
Rehabilitation adherence | 6 months
  Rehabilitation adherence will be measured by the rehabilitation adherence questionnaire which is developed by the research team, and it was validated by stroke and chronic care expert. This scale has 3 items with a 5-point Likert scale, and the score ranges from 3- 15. The higher mean score indicates greater adherence to rehabilitation.
Improved motor function | 6 months
  The motor function will be measured by the Motricity Index (MI) developed by Demeurisse et al. in 1980 which is valid & reliable (α= 0.93) [25]to assess the motor impairment of participants. Three movements for upper (pinch grip, PG; elbow flexion, EF; shoulder abduction, SA) and lower (ankle dorsiflexion, AD; knee extension, KE; hip flexion, HF) limbs are assessed for evaluating motor function. It is a 6-point scale for the arm and leg test; 3 points for trunk control test. A total score ranging from 0 (complete paresis) to 100 (normal strength) and is computed for each limb on both sides, and a side score can be computed by averaging upper and lower limb scores. The higher score indicates better limb function.
Improved self-efficacy | 6 months
  Self-efficacy will be assessed by the generalized self-efficacy scale (GSE) (Jerusalem et al., 1981) [26]. This scale assessed patients' self-efficacy after experiencing post-stroke stress and the strength of an individual's belief in situations. It was translated into the Bengali version and was found valid and reliable (α = 0.7 to 0.91) [27]. It has a total of 10 items with a 4-point Likert scale that ranges from 1= not at all true to 4=exactly true. The lowest score is 10 and the highest score is 40. The higher score indicates better self-efficacy.
Improved emotional status | 6 months
  he emotional status will be assessed using a subdomain of stroke impact scale (SIS) which is valid and reliable for assessing patient-perceived mood, emotional control, and psychological well-being following stroke [28]. This subdomain scale has 9 items with a 5-point Likert scale and score ranges from 9-45. Domain scores will be calculated using standard SIS scoring procedures and transformed to a 0-100 scale, with higher scores indicating less perceived impact of stroke.
Improved participation abilities | 6 months
  Participation ability will be measured by participation/role function subdomain of the stroke impact scale (SIS) to evaluate restrictions in social participation, meaningful activities, and societal roles. This subdomain scale has 8 items with a 5-point Likert scale and score ranges from 8-40. Domain scores will be calculated using standard SIS scoring procedures and transformed to a 0-100 scale, with higher scores indicating less perceived impact of stroke.

CONTACTS AND LOCATIONS:
Overall Officials: Salma Akhter, Principal Investigator — Hiroshima University
Locations (1):
- National Institute of Neuroscience and Hospital, Dhaka, Dhaka Division, Bangladesh

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Feigin VL, Brainin M, Norrving B, Martins SO, Pandian J, Lindsay P, F Grupper M, Rautalin I. World Stroke Organization: Global Stroke Fact Sheet 2025. Int J Stroke. 2025 Feb;20(2):132-144. doi: 10.1177/17474930241308142. Epub 2025 Jan 3. PMID 39635884